CLINICAL TRIAL: NCT07004543
Title: Evaluation of Toe Separators in Foot Health: A Pilot Observational Study (STEP-IN)
Brief Title: Evaluation of Toe Separators in Foot Health
Acronym: STEP-IN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UCV/2023.2024/027.
Record Dates: First submitted 2025-05-09; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Health-Related Behavior
Keywords: Toe separators; Gait analysis; Plantar pressure
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This research follows a single-group pre-post design, also classified as a pre-experimental model. It is a pilot observational study aimed at exploring the initial effects of standard toe separators on foot health in healthy individuals.
  No control group is included, as the main objective is to conduct an early investigation of the biomechanical and physiological impact of these orthotic devices. This design allows the detection of potential trends or preliminary effects, serving as a basis for future, more rigorous studies such as randomized controlled trials.
  Measurements are taken at two time points:
  Pre-intervention: Baseline evaluation without the toe separators.
  Post-intervention: Evaluation after applying the toe separators.
  This model is appropriate for exploratory phases, especially when the phenomenon under investigation-such as the widespread use of standard toe separators-has limited scientific literature and lacks empirical validation.
Who Masked: Outcomes Assessor
Masking Description: Each data set (pre- and post-intervention) will be assigned a random code (e.g., "M1" and "M2") without indicating whether it corresponds to the before or after condition.
  The evaluator responsible for analyzing the results-such as plantar pressures, imaging, or comfort scores-will not have access to the timing or condition of the data. This approach ensures objective interpretation and minimizes potential bias related to expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Toe Separator Intervention (Experimental): Participants in this arm will undergo assessments before and after using standard, non-custom silicone toe separators.
  Interventions: Procedure: Standard Silicone Toe Separator Application
- No-Intervention Control Group (No Intervention): Participants in the control arm will undergo the same evaluation procedures as the intervention group but without the application of toe separators.

INTERVENTIONS:
Procedure: Standard Silicone Toe Separator Application — Participants will be instructed to wear standard, commercially available silicone toe separators during a single evaluation session. The intervention consists of applying the separators between the toes while the participant is barefoot, both in static standing and while walking on a treadmill equipped with a Zebris pressure analysis system. Measurements will be taken immediately before and after the application, including plantar pressure distribution, intermetatarsal spacing (via imaging), digital circulation (via thermography and visual assessment), foot posture (using the Foot Posture Index - FPI-6), and subjective comfort levels (via Visual Analog Scale). The toe separators are not customized and reflect common consumer-grade devices marketed for podiatric or wellness purposes.
  Arms: Standard Toe Separator Intervention

SUMMARY:
This pilot observational study investigates the effects of standard toe separators on foot health in asymptomatic individuals. It aims to evaluate their impact on intermetatarsal spacing, plantar pressure distribution, digital circulation, and user comfort. Through pre- and post-intervention measurements using tools like thermography, gait analysis (Zebris), and the Foot Posture Index, the research seeks to determine whether these commonly used orthotic devices provide measurable benefits or pose risks. The study ultimately contributes to evidence-based podiatric care and public health education.

DETAILED DESCRIPTION:
This research project titled "Evaluation of Toe Separators in Foot Health: A Pilot Observational Study (STEP-IN)" explores the biomechanical and physiological effects of standard, commercially available toe separators on healthy individuals without pre-existing podiatric conditions.

Given the growing popularity of these devices on social media and among the general public-often promoted as tools for correcting deformities, relieving plantar pain, or improving foot posture-this study aims to objectively assess their actual benefits and limitations using scientific methods.

The study employs a pre-post observational design involving 40 adult volunteers. A comprehensive analysis is conducted before and after the application of toe separators, focusing on several key variables:

Intermetatarsal angles and spacing measured through imaging (ultrasound or X-ray).

Gait and plantar pressure distribution assessed with the Zebris system.

Digital circulation evaluated visually and via thermographic imaging.

Foot posture assessed using the validated Foot Posture Index (FPI-6).

Comfort perception measured through a Visual Analog Scale (VAS).

Participants are evaluated during static stance and dynamic walking conditions to determine how the devices affect natural biomechanics. Data is analyzed statistically using SPSS and JASP to compare pre- and post-intervention results, applying appropriate tests based on normality assumptions.

Ethical approval was obtained from the Ethics Committee of the Universidad Católica de Valencia, and all participants provided informed consent.

This project aims not only to inform podiatric practice but also to serve as a foundation for future, larger-scale clinical trials. Additionally, it seeks to counteract misinformation by offering evidence-based insights into a widely used but poorly studied orthotic product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants (without foot pathologies)
* Age 18 or older
* Voluntary participation with signed informed consent
* Students or staff from UCV clinics

Exclusion Criteria:

* Systemic conditions affecting foot sensitivity or circulation (e.g., Raynaud's syndrome,
* Diabetes Type I or II, post-surgical neuralgias, cerebral palsy, acquired hemiplegia, herniated discs with neural involvement, fibromyalgia)
* Presence of any diagnosed podiatric pathology
* Under 18 years of age
* Pregnant individuals
* Inability to understand or sign the informed consent form

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Plantar Pressure Distribution | Baseline and immediately post-intervention
  Zebris treadmill analysis

SECONDARY OUTCOMES:
Intermetatarsal Angles (2nd-3rd, 3rd-4th, 4th-5th) | Baseline and immediately post-intervention
  Imaging (X-ray)
Intermetatarsal Spaces | Baseline and immediately post-intervention
  Quantitative (millimeters)Imaging (X-ray)
Gait Parameters | Baseline and immediately post-intervention
  Zebris gait analysis system
Foot Posture Index | Baseline and immediately post-intervention
  Foot Posture Index (FPI-6).is a clinical tool used to evaluate foot posture in the standing position, taking into account six visual criteria. Each is scored between -2 and +2, giving a total score ranging from -12 (very supinated foot) to +12 (very pronated foot).
  Score range: -12 (maximum supination) to +12 (maximum pronation).
  Interpretation of scores:
  Lower scores indicate a more supinated (less pronated) foot posture. Higher scores indicate a more pronated (less supinated) foot posture.
Perceived Comfort | Baseline and immediately post-intervention
  After the toe separators are applied, the participant will be shown a 10-point Likert-type scale, included in the data collection sheet. It will be explained that they should indicate the degree of comfort they feel while wearing the toe separators by choosing a number from 1 to 10, where:
  1 means very uncomfortable
  10 means very comfortable
  The participant should select the number that best reflects their subjective perception of comfort at that moment.
Digital Circulation | Baseline and immediately post-intervention
  A visual inspection of the participant's feet will be performed to identify any noticeable changes in skin color, swelling, alignment or other external signs of alteration.
Digital Circulation | Baseline and immediately post-intervention
  Thermographic imaging.will be used to assess thermal patterns and skin temperature distribution across the feet. Images will be captured using an infrared thermal camera under standardized environmental conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinicas UCV, Valencia, València, Spain

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be shared through multiple dissemination channels to ensure transparency and accessibility. Upon completion and analysis, findings will be submitted for publication in a peer-reviewed journal specializing in podiatry, biomechanics, or rehabilitation sciences. Additionally, results will be presented at relevant national and international conferences in the fields of podiatry and physical therapy.
Supporting Information: Study Protocol, ICF
Time Frame: All published results and associated materials will be accessible indefinitely through institutional repositories or journal archives,

REFERENCES:
- [Background] Abdalbary SA. Foot Mobilization and Exercise Program Combined with Toe Separator Improves Outcomes in Women with Moderate Hallux Valgus at 1-Year Follow-up A Randomized Clinical Trial. J Am Podiatr Med Assoc. 2018 Nov;108(6):478-486. doi: 10.7547/17-026. Epub 2018 Apr 23. PMID 29683337
- [Background] Dissaneewate T, Na Rungsri T, Cheunchokasan P, Leelasamran W. Comparison between the plantar pressure effects of toe separators and insoles in patients with hallux valgus at a one-month follow-up. Foot Ankle Surg. 2022 Jan;28(1):93-99. doi: 10.1016/j.fas.2021.02.005. Epub 2021 Feb 12. PMID 33612377
- [Background] Krzesniak H, Truszczynska-Baszak A. Toe Separators as a Therapeutic Tool in Physiotherapy-A Systematic Review. J Clin Med. 2024 Dec 19;13(24):7771. doi: 10.3390/jcm13247771. PMID 39768694